CLINICAL TRIAL: NCT04917042
Title: Phase 2 Study Using Tazemetostat in Patients With Recurrent/Refractory and/or Metastatic Malignant Peripheral Nerve Sheath Tumors (MPNST)
Brief Title: Tazemetostat in Malignant Peripheral Nerve Sheath Tumors
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Epizyme, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UF-SC-001; IRB202100865 (Other: UF IRB-01); OCR40197 (Other: University of Florida)
Record Dates: First submitted 2021-06-01; First posted 2021-06-08 (Actual); Results first posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Peripheral Nerve Sheath Tumor
Keywords: metastatic malignant peripheral nerve sheath tumors; Enhancer of zeste homolog 2 (EZH2) inhibition; sarcoma; pediatric; tazemetostat
MeSH Terms: conditions — Nerve Sheath Neoplasms; Neurofibrosarcoma; Inhibition, Psychological; Sarcoma | interventions — tazemetostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- tazemetostat (Experimental)
  Interventions: Drug: Tazemetostat

INTERVENTIONS:
Drug: Tazemetostat — Subjects will receive 520 mg/m2/dose (subjects 12-17 years old) or 800 mg of tazemetostat orally twice daily in 28 day cycles. Subjects will receive treatment with tazemetostat up to 2 years or until disease progression or unacceptable toxicity occurs.
  Other Names: TAZVERIK

SUMMARY:
This phase 2, open label, single arm study will investigate the use of tazemetostat in patients with recurrent/refractory and/or metastatic malignant peripheral nerve sheath tumors.

ELIGIBILITY:
Inclusion Criteria:

* A histologic confirmation of recurrent/refractory and/or metastatic malignant peripheral nerve sheath tumor with Response Evaluation Criteria in Solid Tumors (RECIST) measurable disease
* Patients ≥ 12 years of age at the time of enrollment
* Performance status: 12-15 years old: Lansky > 50; 16-17 years old: Karnofsky > 50; ≥ 18 years old: Eastern Cooperative Group (ECOG) score 0-2
* Subjects must have adequately recovered from the acute toxic effects of all prior anti-cancer therapy per enrolling physician and must meet the following minimum duration from prior anti-cancer directed therapy prior to enrollment.

  * Anti-cancer agents known to be Myelosuppressive: ≥ 28 days after the last dose of agent.
  * Anti-cancer agents not known to be myelosuppressive: > 7 days after the last dose of agent.
  * Antibodies: > 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to Grade < 1.
  * Systemic Corticosteroids: if related to prior therapy > 14 days must have elapsed, or on stable dose for treatment of CNS disease.
  * Hematopoietic growth factors: > 14 days after the last dose of a long-acting growth factor.
  * Interleukins, Interferons, and Cytokines (other than hematopoietic growth factors): > 21 days after the completion of interleukins, interferon or cytokines (other than hematopoietic growth factors).
  * Radiation therapy (XRT)/External Beam Irradiation including Protons: > 14 days after local XRT; > 150 days after traumatic brain injury, craniospinal XRT or if radiation to > 50% of the pelvis; > 42 days if other substantial bone marow radiation.
  * Radiopharmaceutical therapy: > 42 days after systemically administered radiopharmaceutical therapy.
  * Major surgery > 14 days prior, with evidence of wound healing and no active surgical complications
* Subjects must not have had prior exposure to Tazemetostat or other inhibitor(s) of EZH2
* Adequate laboratory values of organ function, defined as:

  * Peripheral absolute neutrophil count (ANC) > 1000/mm3.
  * Platelet count > 100,000/mm2 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment).
  * Hemoglobin > 8.0 g/dL at baseline (may receive RBC transfusions).
  * Creatinine clearance or radioisotope GFR > 70 ml/min/1.73 m2, or serum creatinine based on age/gender
  * Total bilirubin < 1.5 ULN or direct bilirubin < 1 x ULN.
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 x ULN; if liver metastases present, then AST and ALT must be < 5 x ULN.
  * Serum albumin > 2 g/dL.
  * Coagulation INR < 1.5, while on anti-coagulation INR < 2.5.
* Nervous system disorders (CTCAE v5.0) resulting from prior therapy must be < Grade 2, with the exception of decreased tendon reflex (DTR). Any grade of DTR is eligible.
* Subjects must not have more than one active malignancy at the time of enrollment
* Written informed consent obtained from the subject and the subject agrees to comply with all the study-related procedures. All subjects and/or their parents or legally authorized representatives must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional standard practice.
* Use of contraception:

  * Women of childbearing potential (WOCBP) who are heterosexually active must be using two highly effective methods of contraception to avoid pregnancy throughout the study and for at least 6 months after the last dose of study drug to minimize the risk of pregnancy as Tazemetostat might counteract the effects of hormonal contraceptives. Birth control methods that can be used while in this study include: established use of oral, injected or implanted hormonal birth control or placement of an intrauterine device [IUD] or intrauterine system [IUS]. They or their partner must also use a second method, (e.g., condom with spermicidal foam/gel/film/cream/suppository or occlusive cap [diaphragm or cervical/vault caps] with spermicidal foam/gel/film/cream/suppository. If their male partner is vasectomized, they do not need to use any of the birth control methods listed above. The type of birth control they use must be discussed with the study doctor before beginning the study. The study doctor must approve the method you use before they can enter the study. Prior to study enrollment, women of childbearing potential must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy.
  * Males with female partners of child-bearing potential must agree to use physician-approved contraceptive methods (e.g., abstinence, condoms,vasectomy) throughout the study and should avoid donating sperm, for 90 days following the last dose of study drug.

Exclusion Criteria:

* Subjects who are currently taking the following concomitant medications:

  * Anti-cancer Agents: Subjects who are currently receiving other anti-cancer agents are not eligible.
  * CYP3A4 Agents: Subjects who are currently receiving drugs that are strong inducers or strong inhibitors of CYP3A4 are not eligible. Strong inducers or inhibitors of CYP3A4 are prohibited from 14 days prior to the first dose of Tazemetostat to the end of the study. Note: Dexamethasone for CNS tumors or metastases, on a stable dose, is allowed.
  * Grapefruit, grapefruit juice, Seville oranges and food/drinks containing them should be avoided one week before the first dose of the study intervention
* Subjects who are acutely ill with an uncontrolled active infection on systemic anti-infective agents are not eligible.
* Subjects with a prior history of T-cell lymphoblastic lymphoma/T-cell acute lymphoblastic leukemia, myelodysplastic syndrome (MDS), acute myeloid leukemia (AML), B-cell acute lymphoblastic leukemia (B-ALL) or other myeloproliferative neoplasm (MPN).
* Subjects who have any of the following underlying major cardiac issues or conditions:

  * Known QTc prolongation or documentation
  * Documented New York Heart Association (NYHA) Class III or IV congestive heart failure.
  * Myocardial infarction within 6 months prior to registration.
  * Unstable angina within 6 months prior to registration.
  * Symptomatic arrhythmia.
* Subjects who in the opinion of the investigator may be high risk for treatment complications or unable to comply with the safety monitoring requirements of the study
* Heterosexually active males or females of reproductive potential may not participate unless they have agreed to use two highly effective contraceptive methods for the duration of study treatment as Tazemetostat might counteract the effects of hormonal contraceptives. Female subjects of childbearing potential should agree to remain abstinent or use adequate contraceptive methods for 6 months after the last dose of Tazemetostat. Male subjects should agree to remain abstinent or use adequate contraceptive methods, and agree to refrain from donating sperm, and for 90 days after the last dose of Tazemetostat.
* Females who are pregnant or breastfeeding will not be entered on this study because there is currently no available information regarding human fetal or teratogenic toxicities. Pregnancy tests must be obtained in girls who are post-menarchal.
* Administration of a vaccine containing live virus within 30 days prior to the first dose of trial treatment. Note: Most flu vaccines are killed viruses, with the exception of the intra-nasal vainer (Flu-Mist) which is an attenuated live virus and therefore prohibited for 30 days prior to first dose. Non-live versions of the COVID-19 vaccine are allowed.
* Prisoners or subjects who are involuntarily incarcerated, or subjects who are compulsorily detained for treatment of either a psychiatric or physical illness.
* Known hypersensitivity to tazmetostat or any component of the formulation of tazemetostat
* Inability to take oral medication OR have malabsorption syndrome or any other uncontrolled gastrointestinal condition (eg, nausea, diarrhea, vomiting) that might impair the bioavailability of tazmetostat

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2026-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Lagmay, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tazemetostat
Started | 10
Completed | 9
Not Completed | 1
Not completed — Subject is still on long-term follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tazemetostat
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 40 [20 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Assess the objective response rate, defined as the proportion of subjects who achieve either a complete response or partial response based on radiographic evaluation of treatment response via RECIST1.1. A complete response is the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. A partial response is at least a 30% decrease in the sum of diameter of target lesions, taking as reference the baseline sum diameters.
Time Frame: 143 days
Population: One participant was not evaluable for this outcome measure because a RECIST response was not obtained after baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Tazemetostat
Number analyzed (Participants) | 9
percentage of participants | 0

2. Secondary Outcome: Progression Free Survival
Description: Determine the progression free survival, defined as the length of time from the date of start of treatment to the date of disease progression per RECIST 1.1 criteria. Per RECIST 1.1 criteria, disease progression is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (including the baseline sum if that is the smallest). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of 1 or more new lesions is also considered progression.
Time Frame: 143 days
Population: One participant was not evaluable for this outcome measure because a RECIST response was not obtained after baseline.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tazemetostat
Number analyzed (Participants) | 9
months | 1.9 [1.2 to NA] — The upper limit of the confidence interval is not estimable because fewer than half of the participants had progressed by the end of follow-up.

3. Secondary Outcome: Time to Progression
Description: Determine the time to progression, defined as the length of time from the start of treatment until disease progression by RECIST 1.1 criteria. Per RECIST 1.1 criteria, disease progression is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (including the baseline sum if that is the smallest). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of 1 or more new lesions is also considered progression.
Time Frame: 143 days
Population: One participant was not evaluable for this outcome measure because a RECIST response was not obtained after baseline.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tazemetostat
Number analyzed (Participants) | 9
months | 1.9 [1.2 to NA] — The upper limit of the confidence interval is not estimable because fewer than half of the participants had progressed by the end of follow-up.

4. Secondary Outcome: Clinical Benefit
Description: Determine the clinical benefit using the Numbered Pain Rating Scale. For this scale, the subject rates their pain on a scale of 0 to 10. Zero means "no pain," and 10 means "the worst possible pain." For each patient, the mean pain rating scale score was computed by adding all the non-missing scores the patient had and then taking the average.
Time Frame: 143 days
Population: One participant was not included as they were not evaluable.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tazemetostat
Number analyzed (Participants) | 9
score on a scale | 3.4 (2.7)

5. Secondary Outcome: Clinical Benefit Rate
Description: Assess the clinical benefit rate, defined as the proportion of subjects with complete or partial response or stable disease (by RECIST 1.1 criteria) lasting at least 4 months.
  Per RECiST 1.1 criteria, a complete response is the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. A partial response is at least a 30% decrease in the sum of diameter of target lesions, taking as reference the baseline sum diameters. Stable disease is defined as having neither sufficient shrinkage for a partial response nor sufficient increase for progressive disease, taking as reference the smallest sum diameters while on study.
Time Frame: 143 days
Population: One participant was not evaluable for this outcome measure because a RECIST response was not obtained after baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Tazemetostat
Number analyzed (Participants) | 9
percentage of participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the start of study therapy until 28 days after the last dose of study treatment. Adverse events were collected for up to 169 days.
Description: Adverse events were assessed by the principal investigator, the treating sub-investigator, and/or the study coordinator from the start of study therapy until 28 days after the last dose of study treatment. Adverse events were assessed by physical examination, labs, and subject self-reports.
Arm/Group | Tazemetostat
All-Cause Mortality (participants affected / at risk) | 9/10
Serious Adverse Events (participants affected / at risk) | 4/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tazemetostat (N=10)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Superior vena cava syndrome (Vascular disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 1
Lung infection (Infections and infestations) | 1
Disease Progression (General disorders) | 1
Progressive Disease (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tazemetostat (N=10)
Anal fissure (Gastrointestinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 1
Anxiety (Psychiatric disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Blood bilirubin increased (Investigations) | 1
Chest pain (Musculoskeletal and connective tissue disorders) | 1
Cholesterol high (Investigations) | 1
Constipation (Gastrointestinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Depression (Psychiatric disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Dysuria (Renal and urinary disorders) | 1
Fatigue (General disorders) | 6
Flu-like symptoms (General disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Hallucinations (Psychiatric disorders) | 1
Hot flashes (Vascular disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Insomnia (Psychiatric disorders) | 1
Lethargy (Nervous system disorders) | 1
Lymphocyte count decreased (Investigations) | 1
Memory impairment (Nervous system disorders) | 1
Movements involuntary (Nervous system disorders) | 1
Muscle cramp (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 7
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 2
Pruritis (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 2
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1
Sinus tachycardia (Cardiac disorders) | 2
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Vomiting (Gastrointestinal disorders) | 5
Weight loss (Investigations) | 1
Wound infection (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-12): https://cdn.clinicaltrials.gov/large-docs/42/NCT04917042/Prot_SAP_000.pdf